CLINICAL TRIAL: NCT00003926
Title: A Phase I Study of the Chemoprotectant Amifostine With Autologous Stem Cell Transplantation for High Risk or Relapsed Pediatric Solid Tumors and Brain Tumors
Brief Title: Amifostine to Protect From Side Effects of PSCT in Treating Patients With Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Withdrawn due to slow accrual
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: John Perentesis, MD, Masonic Cancer Center, University of Minnesota
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1997LS053; UMN-MT-9713 (Other: Blood and Marrow Transplantation Program); UMN-9712M00074 (Other: IRB, University of Minnesota)
Record Dates: First submitted 1999-11-01; First posted 2003-05-02 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Brain and Central Nervous System Tumors; Childhood Germ Cell Tumor; Chordoma; Kidney Cancer; Liver Cancer; Neuroblastoma; Ovarian Cancer; Retinoblastoma; Sarcoma
Keywords: soft tissue sarcoma; regional neuroblastoma; disseminated neuroblastoma; recurrent Wilms tumor; recurrent retinoblastoma; recurrent adult brain tumor; adult rhabdomyosarcoma; ovarian germ cell tumor; chordoma; ovarian sarcoma; unresectable neuroblastoma; desmoplastic small round cell tumor; rhabdomyosarcoma; Ewing sarcoma; neuroectodermal tumor; teratoma; malignant testicular germ cell tumor; malignant ovarian germ cell tumor; extragonadal germ cell tumor; malignant germ cell tumor; hepatoblastoma; liver cancer; medulloblastoma; cerebellar astrocytoma; brain stem glioma; glioma; cerebral astrocytoma; ependymoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Chordoma; Kidney Neoplasms; Liver Neoplasms; Neuroblastoma; Ovarian Neoplasms; Retinoblastoma; Sarcoma; Wilms Tumor; Brain Neoplasms; Rhabdomyosarcoma; Desmoplastic Small Round Cell Tumor; Sarcoma, Ewing; Neuroectodermal Tumors; Teratoma; Testicular Neoplasms; Ovarian Germ Cell Cancer; Hepatoblastoma; Medulloblastoma; Glioma; Astrocytoma; Ependymoma | interventions — Amifostine; Busulfan; Filgrastim; Granulocyte Colony-Stimulating Factor; Melphalan; Thiotepa; Peripheral Blood Stem Cell Transplantation; Bone Marrow Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Solid/brain tumor patients (1-18 years) (Experimental): Patients with solid tumor or brain tumor in the 1-18 years old stratum.
  Interventions: Drug: amifostine trihydrate; Drug: busulfan; Drug: filgrastim; Drug: melphalan; Drug: thiotepa; Procedure: peripheral blood stem cell transplantation (PBSC)
- Solid/brain tumor patients (19-45 years) (Experimental): Patients with solid tumor or brain tumor in the 19-45 years old stratum.
  Interventions: Drug: amifostine trihydrate; Drug: busulfan; Drug: filgrastim; Drug: melphalan; Drug: thiotepa; Procedure: peripheral blood stem cell transplantation (PBSC)

INTERVENTIONS:
Drug: amifostine trihydrate — Patients receive amifostine intravenous (IV) over 5 minutes beginning 30 minutes prior to melphalan and thiotepa administration on days -5 to -1.
  Cohorts of 3-6 patients receive escalating doses of amifostine until the maximum tolerated dose is determined.
  Other Names: Ethyol
Drug: busulfan — Patients receive oral busulfan every 6 hours on days -8 to -6.
  Other Names: Busulfex
Drug: filgrastim — All patients receive filgrastim (G-CSF) IV for 1 week.
  Other Names: granulocyte colony-stimulating factor; G-CSF
Drug: melphalan — melphalan intravenous (IV) over 30 minutes on days -5 and -4
  Other Names: Alkeran
Drug: thiotepa — thiotepa intravenous (IV) over 2 hours on days -3 and -2.
  Other Names: Thioplex
Procedure: peripheral blood stem cell transplantation (PBSC) — PBSC are reinfused on day 0
  Other Names: bone marrow transplant

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells. Chemoprotective drugs such as amifostine may protect normal cells from the side effects of high-dose chemotherapy.

PURPOSE: Phase I trial to study the effectiveness of amifostine in protecting from the side effects of peripheral stem cell transplantation in treating patients who have high-risk or relapsed solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the dose-limiting toxicity of amifostine chemoprotection with peripheral blood stem cell transplantation plus chemotherapy in patients with high-risk or relapsed solid tumors or brain tumors.
* Determine response or time to disease progression in patients treated with this regimen.

OUTLINE: This is a dose-escalation study of amifostine. Patients are stratified according to age (1 to 18 vs 19 to 45 years).

All patients receive filgrastim (G-CSF) IV for 1 week. On day 6 of G-CSF administration, patients undergo peripheral blood stem cell (PBSC) harvest followed by chemotherapy.

Patients receive oral busulfan every 6 hours on days -8 to -6 followed by melphalan IV over 30 minutes on days -5 and -4 and thiotepa IV over 2 hours on days -3 and -2. Patients receive amifostine IV over 5 minutes beginning 30 minutes prior to melphalan and thiotepa administration on days -5 to -1. PBSC are reinfused on day 0.

Cohorts of 3-6 patients receive escalating doses of amifostine until the maximum tolerated dose is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed on day 50; at 3, 6, and 9 months; and at 1, 2, and 3 years post PBSC transplantation.

PROJECTED ACCRUAL: A maximum of 60 patients (30 per stratum) will be accrued for this study within 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed high-risk or relapsed solid tumors or brain tumors, including:

  * Metastatic or relapsed Ewing's sarcoma
  * Metastatic or relapsed rhabdomyosarcoma
  * Refractory Wilms' tumor
  * Diffuse anaplastic Wilms' tumor
  * Stage III or IV neuroblastoma
  * Recurrent retinoblastoma
  * Metastatic or relapsed germ cell tumors
  * Metastatic or relapsed other soft tissue sarcomas
  * Small cell ovarian sarcoma
  * Metastatic or relapsed primitive neuroectodermal tumors of the bone
  * Recurrent brain tumors
  * Desmoplastic small round cell tumors
  * Recurrent or metastatic chordomas
  * Metastatic or relapsed hepatoblastoma
* Patients receive peripheral blood stem cell transplantation only if in complete remission or in very good partial remission with no disease progression
* Must have radiologic, nuclear image, or histologic verification of relapse
* Age 1 to 45
* Performance status:Karnofsky 70-100%
* Absolute neutrophil count greater than 1,000/mm^3
* Platelet count greater than 100,000/mm^3
* Hemoglobin count at least 10 g/dL
* Bilirubin less than 2 times upper limit of normal (ULN)
* SGOT or SGPT less than 2.5 times ULN
* Creatinine less than 2 times ULN
* Creatinine clearance greater than 70 mL/min
* Cardiac shortening fraction greater than 30%
* Cardiac ejection fraction greater than 45%
* At least 1 week since prior hematopoietic growth factor and recovered
* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas) and recovered
* Recovered from any prior therapy

Exclusion Criteria:

* Osteogenic sarcoma
* Less than 4 months
* Uncontrolled bleeding
* Congestive heart failure
* Uncontrolled hypertension
* Asthma
* Pregnant or nursing
* Uncontrolled metabolic disease
* Active severe infection
* Allergy to aminothiol compounds
* Prior bone marrow transplantation
* Other concurrent investigational agents

Ages: 1 Year to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 1998-11; Primary Completion 2002-08 (Actual); Study Completion 2003-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John P. Perentesis, MD, Study Chair — Masonic Cancer Center, University of Minnesota
Locations (1):
- University of Minnesota Cancer Center, Minneapolis, Minnesota, United States